CLINICAL TRIAL: NCT01293877
Title: Laparoscopic Gastric Plication for Treatment of Morbid Obesity
Brief Title: Laparoscopic Gastric Plication Compared With Laparoscopic Sleeve Gastrectomy
Acronym: LGP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bikkur Holim Hospital (Other)
Responsible Party: Sergio Susmallian, Bikkur Holim Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GP111BH
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Morbid Obesity
Keywords: Laparoscopy; obesity; gastric; restrictive
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LGP (Other): Patient underwent surgery for morbid obesity treatment between 18 to 60 years, and BMI of 40 ore more will divided in two groups, one hundred will be schedule for laparoscopic gastric plication. Our theory for this arm is that the procedure can offer the same results than the second arm with less cost and safety, reversibility included.
  Interventions: Procedure: Laparoscopy surgery for morbid obesity
- LSG (Other): The patients in a total of one hundred will be schedule for laparoscopic sleeve gastrectomy. The is our control for development of the study.
  Interventions: Procedure: Laparoscopy surgery for morbid obesity

INTERVENTIONS:
Procedure: Laparoscopy surgery for morbid obesity — The intervention will compare the 2 restrictive procedures one sleeve gastrectomy and gastric plication/

SUMMARY:
The study must be performed in 100 patients suffering from morbid obesity, the procedure will be performed under general anesthesia doing two or three layers of suture to achieves gastric imbrication until transform the stomach to a sleeve. The patients will be followed during the time for 6 month, 1 year, two years and 5 years.

DETAILED DESCRIPTION:
The patients will be selected with BMI more than 40, the operation will be primary between 18 to 60 years old. The patients will be informed about the procedure and different options. The patients will be in admission board for two or three days and any event will be recorded. the follow up will be recorded by the nurse, the surgeon and the dietitian, laboratory parameter includes CBC, T4,T3, TSH, ferrum, transferrin, ferritin, vit. B12, SMA, lipids, The end point will be the EBW achieved and events occurred.

ELIGIBILITY:
Inclusion Criteria:

* BMI 40 or more
* Age between 18-60 years old
* ASA score 1-2

Exclusion Criteria:

* BMI less than 40
* Severe illness
* Psychiatric disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Body Mass index loss | 6mont.
  The body mass index will be compared before the procedure and after at time frames.

SECONDARY OUTCOMES:
Complications Quality of life | 6 month
  complications compared one with the second procedure, qol, possibility to eat.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio g Susmallian, dr, Principal Investigator
Locations (1):
- Bikur Holim Hospital, Jerusalem, Jerusalem, Israel